CLINICAL TRIAL: NCT06462326
Title: A Phase 1, Randomized, Double-Blind Study to Compare the Effect of Omadacycline PO Versus Moxifloxacin PO on the Gut Microbiota in Healthy Adult Volunteers
Brief Title: A Study to Compare the Effect of Omadacycline Versus Moxifloxacin in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zai Lab (Hong Kong), Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: ZL-2401-005
Record Dates: First submitted 2024-04-29; First posted 2024-06-17 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Moxifloxacin; omadacycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moxifloxacin (Active Comparator): Moxifloxacin PO (400 mg)q24h D1-D10
  Interventions: Drug: Moxifloxacin Oral Tablet
- Omadacycline (Experimental): Omadacycline PO (450 mg) q24h D1-D2 PO (300 mg) q24h D3-D10
  Interventions: Drug: Omadacycline Oral Tablet

INTERVENTIONS:
Drug: Moxifloxacin Oral Tablet — 400mg per tablet
  Other Names: Avelox
  Arms: Moxifloxacin
Drug: Omadacycline Oral Tablet — 150 mg per tablet
  Other Names: NUZYRA
  Arms: Omadacycline

SUMMARY:
This is a randomized (1:1), double-blind, double-dummy, phase I study to compare the effects of Omadacycline versus Moxifloxacin on gut microbiota and the resistomes in healthy adult volunteers.The study consists of 3 phases: Screening, double-blind treatment, and follow-up. Healthy volunteers aged 18-40 years, who meet entry criteria, are randomly assigned to a treatment group using an Interactive Voice Response System/Interactive Web Response System (IxRS) and receive the first dose of the study drug.

DETAILED DESCRIPTION:
The study consists of 3 phases: Screening, double-blind treatment, and follow-up. Healthy volunteers aged 18-40 years, who meet entry criteria, are randomly assigned to a treatment group using an Interactive Voice Response System/Interactive Web Response System (IxRS) and receive the first dose of the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an Informed Consent Form (ICF) prior to the commencement of any study-related procedures.
2. Chinese healthy male and female subjects aged between 18 and 40 years (inclusive).
3. Body mass index (BMI) between 18.5 and 23.9 kg/m2 (inclusive).
4. Complete the stool sample collections required during screening.

Exclusion Criteria:

1. Subjects with clinically significant medical history of cardiovascular, hepatic, renal, gastrointestinal or psychiatric conditions, or any other condition as deemed by the investigators that may potentially jeopardize subject safety or impact study outcomes.
2. Subjects who have undergone any major surgery within 4 weeks prior to the first dose of study drug administration.
3. Subjects who have previously undergone gastrointestinal surgery that may affect the absorption of the study drug (eg. Intestinal resection surgery, fistula surgery).
4. During screening, subjects with positive tests for hepatitis C antibodies, hepatitis B surface antigen, or hepatitis B virus (HBV) DNA or HBV RNA, or known positive tests for human immunodeficiency virus (HIV).
5. Subjects with Fridericia-corrected QT interval (QTcF) > 450 milliseconds (males) or > 470 milliseconds (females); or known to have long QT syndrome; or using medications that may cause arrhythmia or prolong QT interval, and/or experiencing tachyarrhythmia.
6. Subjects with a history of irritable bowel syndrome (with or without constipation) -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
Changes in the types of microbial resistomes. | 3months
  Metagenome will be extracted from fecal samples of ME population and subjected to second-generation high-throughput sequencing. Bioinformatics will be employed to study the changes in the types of resistance-related genes of microbiota during the drug administration process in the microbiologically evaluable population. This outcome is based on second-generation high-throughput sequencing. the outcome is to test the genes to confirm the changes in types of microbial resistors in different stages.
Changes in the quantity of microbial resistomes. | 3months
  Metagenome will be extracted from fecal samples of ME population and subjected to second-generation high-throughput sequencing. Bioinformatics will be employed to study the changes in the quantity of resistance-related genes of microbiota during the drug administration process in the microbiologically evaluable population.This outcome is based on second-generation high-throughput sequencing. the outcome is to test the gene to confirm the changes in quantity of microbial resistors in different stages .
Changes in the abundance of microbial resistomes. | 3months
  Metagenome will be extracted from fecal samples of ME population and subjected to second-generation high-throughput sequencing. Bioinformatics will be employed to study the changes in the abundance of resistance-related genes of microbiota during the drug administration process in the microbiologically evaluable population.This outcome is based on second-generation high-throughput sequencing. the outcome is to test the genes to confirm the changes in abundance of microbial resistors in different stages.

SECONDARY OUTCOMES:
Changes in the microbial composition | 3months
  Metagenome will be extracted from fecal samples of ME population and subjected to second-generation high-throughput sequencing. Principal component analysis will be employed to study the changes in the structure of microbiota during the drug administration process in the microbiologically evaluable population. This outcome is based on the result of principal component analysis to confirm the microbial composition in different stages based on different genes.
Changes in the microbial functionality | 3months
  Metagenome will be extracted from fecal samples of ME population and subjected to second-generation high-throughput sequencing. Principal coordinates analysis will be employed to study the changes in the structure of microbiota during the drug administration process in the microbiologically evaluable population. This outcome is based on result of principal coordinates analysis to confirm the microbial functionality in different stages based on different genes.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Liu, Principal Investigator — Zhejiang University; Yonghong Xiao, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, China